CLINICAL TRIAL: NCT03146650
Title: Phase II Study of Nivolumab and Ipilimumab for Treatment of Metastatic/Recurrent Adenoid Cystic Carcinoma of All Anatomic Sites of Origin and Non-adenoid Cystic Carcinoma Malignant Tumors of the Salivary Gland
Brief Title: Nivolumab and Ipilimumab in Treating Patients With Metastatic/Recurrent ACC of All Sites and Non-ACC Salivary Gland Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16N03; STU00204579 (CTRP (Clinical Trial Reporting Program)); NU 16N03 (Other: Northwestern University); P30CA060553 (NIH); NCI-2017-00406 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Major Salivary Gland Carcinoma; Minor Salivary Gland Carcinoma; Recurrent Salivary Gland Carcinoma; Stage IV Major Salivary Gland Carcinoma; Stage IVA Major Salivary Gland Carcinoma; Stage IVB Major Salivary Gland Carcinoma; Stage IVC Major Salivary Gland Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1, 15, 29, 43, 57, and 71 of course 1 and on days 1 and 15 of course 2, over 60 minutes on days 29 and 57 of course 2 and on days 1, 29, and 57 of subsequent courses. Patients also receive ipilimumab over 90 minutes on days 1 and 43. Courses repeat every 84 days in the absence of disease progression or unexpected toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies the efficacy (the effect on the tumor) and the safety (the effect on the body) of the study drugs when given as a combination in participants with this type of cancer. Another purpose of the study is to see which tumor markers (proteins in the blood that the body produces in response to the cancer) lead to better results in participants treated with the study drugs. Nivolumab and ipilimumab are antibodies, which are human proteins that recognize and attach to a part of the tumor and/or body's immune cells. They work in slightly different ways to activate the immune system and help the body's immune system to work against tumor cells. Nivolumab and ipilimumab are investigational because they are not approved by the FDA to be used for the type of cancer being studied.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess median progression-free survival rate (PFSR) as well as PFSR at 6 and 12 months in patients with recurrent or metastatic adenoid cystic carcinoma (ACC) treated with a combination of nivolumab and ipilimumab.

SECONDARY OBJECTIVES:

I. To assess the efficacy of nivolumab and ipilimumab according to response rate (RR), disease control rate (DCR; complete response [CR], partial response [PR], and stable disease [SD] at 6 and 12 months), overall survival (OS) and progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with recurrent or metastatic ACC.

II. To assess the efficacy of nivolumab and ipilimumab according to overall response rate (ORR), DCR, progression free survival (PFS), and OS in patients with recurrent or metastatic ACC using immune-related response criteria (irRC) criteria.

III. To assess the safety and tolerability profile of nivolumab and ipilimumab therapy in patients with recurrent or metastatic ACC using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

TERTIARY OBJECTIVES:

I. Assess safety, tolerability and activity of Nivolumab and Ipilimumab in non-ACC malignant salivary gland tumors (MSGT's) using clinical benefit rate (CBR), ORR, PFS, OS.

II. To assess the predictive value of genomic aberrations observed upon comprehensive genomic profiling of the tumor deoxyribonucleic acid (DNA) derived from archival tumor tissue, if available, or blood from patients with recurrent or metastatic ACC and non-ACC MSGTs.

III. Circulating cell free DNA genomic profiling will also be performed at baseline and during treatment with each imaging to explore the genomic landscape of clonal evolution that may elucidate mechanisms behind response or resistance with immunotherapy in adenoid cystic carcinoma and non-ACC MSGTs.

IV. Correlation between expression of PD-L1 and response to treatment will be explored in all patients enrolled in the study.

V. Correlations between other markers of inflammatory/immune signature will be performed that may include but not be limited to PD-1, OX40, CD73, CD39, T cell immunoglobulin and mucin domain containing protein 3 (TIM3), GITRL, CTLA-4, CD3, CD4, CD8, protein tyrosine phosphatase receptor type C (CD45RO), forkhead box P3 (FOXP3), and granzyme by immunohistochemistry analysis and/or flow cytometry.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on days 1, 15, 29, 43, 57, and 71 of course 1 and on days 1 and 15 of course 2, over 60 minutes on days 29 and 57 of course 2 and on days 1, 29, and 57 of subsequent courses. Patients also receive ipilimumab over 90 minutes on days 1 and 43. Courses repeat every 84 days in the absence of disease progression, unexpected toxicity, or withdrawal of consent.

After completion of study treatment, patients are followed up for 30 days, every 4 weeks for 12 weeks, and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic/recurrent adenoid cystic carcinoma (ACC) or non-adenoid cystic carcinomas (non-ACC) of major or minor salivary glands
* Patients must have evidence of disease progression and cannot be a candidate for surgical treatment

  * NOTE: Disease progression is defined as one of the following occurring within the 6 months prior to study entry:

    * At least a 20% increase in radiologically or clinically measurable lesions
    * Appearance of any new lesions or
    * Symptomatic and/or deterioration in clinical status
* Patients must have received at least one prior line of systemic therapy

  * NOTE: There is no limit to the number of prior therapies for stage IV disease
  * NOTE: Patients should not be a candidate for surgical treatment
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v1.1
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) status of 0-2

  * NOTE: ECOG performance status 3 will be allowed only if thought to be directly secondary to adenoid cystic carcinoma disease by treating physician
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: leukocytes >= 2,000/mcL
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: absolute neutrophil count >= 1,500/mcL, regardless of transfusion or growth factor support
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: platelets >= 100,000/mcl, regardless of transfusion or growth factor support
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: total bilirubin total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome or liver metastasis, who can have total bilirubin < 3.0 x ULN)
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN) (or =< 5 times ULN in case of liver metastasis)
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined by: serum creatinine of < 3.0 X ULN (upper limit of normal) or creatinine clearance > 30 mL/minute (using Cockcroft/Gault formula)
* Patients with history of central nervous system (CNS) metastases are eligible if CNS disease has been stable for at least 6 weeks prior to study registration in the opinion of the investigator and does not require corticosteroids (of any dose) for symptomatic management

  * NOTE: Only patients with a known history or indication of CNS disease are required to have CNS imaging prior to study entry
* Females of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours of registration

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP and men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and the designated post-treatment period
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients must not have had chemotherapy or radiotherapy =< 28 days prior to study registration
* Patients who have not recovered to =< grade 1 or tolerable grade 2 from adverse events due to agents administered >= 28 days earlier are not eligible
* Patient must not be a candidate for surgical treatment or radiation
* Patients may not be receiving any other investigational agents =< 28 days prior to registration
* Patients who have had prior exposure to immune checkpoint inhibitors are not eligible; please contact principal investigator, 312-926-4248 for specific questions on potential interactions

  * NOTE: Immune checkpoint inhibitors working through OX40 are an exception (for example, MEDI6383, MEDI6469, MEDI0562, oxelumab, and PF-04518600) and are permitted >= 28 days prior to study registration
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as SLE
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome
  * NOTE: Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection (including minor localized infections) requiring oral or IV treatment
  * Symptomatic class 3 or 4 congestive heart failure, defined as a clinical syndrome resulting from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill with or eject blood
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients should not have any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug

  * NOTE: Inhaled or topical steroids and adrenal replacement steroids at any dose are permitted in the absence of active autoimmune disease; a brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Female patients who are pregnant or nursing are not eligible
* No other prior malignancy is allowed except for the following:

  * Adequately treated basal cell or squamous cell skin cancer,
  * In situ cervical cancer,
  * Or any other cancer from which the patient has been disease free for at least three years
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) is not permitted
* Any known positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection is not permitted
* Patients who received a live, attenuated vaccine =< 30 days before study registration or are anticipated to require such a live attenuated vaccine are not eligible

  * NOTE: Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine (e.g., FluMist) =< 30 days prior to study registration or at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2025-08-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Matsangou, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Chae YK, Duan R, Chung LI, Oh Y, Alexiev B, Shin S, Kim S, Helenowski I, Matsangou M, Villaflor V, Mahalingam D. Phase II Study of Nivolumab and Ipilimumab for Treatment of Metastatic/Recurrent Adenoid Cystic Carcinoma (ACC) of all Anatomic Sites of Origin and Other Malignant Salivary Gland Tumors. Cancer Med. 2025 Apr;14(7):e70724. doi: 10.1002/cam4.70724. PMID 40166913
- [Derived] Tchekmedyian V. Salivary Gland Cancers. Hematol Oncol Clin North Am. 2021 Oct;35(5):973-990. doi: 10.1016/j.hoc.2021.05.011. PMID 34503735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened for accrual on May 19, 2017 with goal of 63 patients. The first patient started treatment June 12, 2017. The study closed Aug. 9, 2019 without meeting the total accrual goal due to the pharma company deciding to close the study.
Groups:
- Nivolumab + Ipilimumab: Nivolumab and ipilimumab combination will be administered intravenously until disease progression or intolerable toxicity.
  Nivolumab: Given at 240mg over 30 minutes (-5 / +15 minutes) every 2 weeks starting with Cycle 1 Day 1 for the first 16 weeks (1 cycle = 12 weeks). Starting with Cycle 2 Day 29, nivolumab will be given at 480mg IV over 60 minutes (-10 / +15 minutes) every 4 weeks.
  Ipilimumab: Given at 1mg/Kg every 6 weeks starting with Cycle 1 Day 1 over approximately 90 minutes (-5 / +15 minutes).
  On days when both nivolumab and ipilimumab are administered, nivolumab should be given first, followed by ipilimumab about 30 minutes after completion of nivolumab.
  Patients will be assessed for response every 12 weeks (±7 days).
Period: Registered for Study
Arm/Group | Nivolumab + Ipilimumab
Started | 25
Received First Dose of Study Drug | 24
Completed | 24
Not Completed | 1
Not completed — Did not continue to meet protocol eligibility criteria after registration. | 1
Period: Completed Cycle 1 of Treatment(Nivo+Ipi)
Arm/Group | Nivolumab + Ipilimumab
Started | 24
Completed | 23
Not Completed | 1
Not completed — Adverse Event | 1
Period: Continued to Cycle 2 and Beyond
Arm/Group | Nivolumab + Ipilimumab
Started (Nivolumab and ipilimumab administered intravenously until disease progression/intolerable toxicity.) | 23
Reached First Response Assessment | 23
Received Cycle 2 Dose of Study Drugs | 21
Completed (2 patients discontinued after completing Cycle 1 due to disease progression.) | 19
Not Completed | 4
Not completed — Still on treatment | 2
Not completed — Progressive Disease | 2
Period: 2 Year Follow-up
Arm/Group | Nivolumab + Ipilimumab
Started (Patients who received one dose of study drug and have discontinued treatment go into follow-up.) | 22
Completed | 3
Not Completed | 19
Not completed — Death | 11
Not completed — Still in follow-up | 7
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Only patients who received at least one dose of study drug are included in the demographics section.
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
adenoid cystic carcinoma vs non-adenoid cystic carcinoma [Count of Participants; unit: Participants]
  Adenoid Cystic Carcinoma | 19
  Non-Adenoid Cystic Carcinoma | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-Free Survival assessed per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria at time of first study treatment. PFS defined as absence of death and of progressive disease. Progressive disease per RECIST v. 1.1 defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). The appearance of one or more new lesions is also considered progression. Response rates and 95% confidence intervals will be calculated using exact binomial probability distributions for discrete outcomes. Efficacy will be evaluated in all patients who receive at least one dose of study treatment and have had their disease re-evaluated.
Time Frame: From the start of treatment and every 12 weeks during treatment, for up to two years, where 1 cycle =12 weeks/84 days, and range of cycles attempted was 1-11.
Population: Patients with recurrent or metastatic Adenoid cystic carcinoma (ACC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 19
percentage of participants
  progression free survival (12 months) | 47.37 [29.49 to 76.09]
  progression free survival (6 months) | 63.16 [44.8 to 89.04]

2. Primary Outcome: Median Progression-free Survival
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Patients with adenoid cystic carcinoma only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 19
months | 8.28 [5.49 to 27.99]

3. Secondary Outcome: Response Rate (RR)
Description: Response rate (RR) is percentage of patients whose cancer shrinks or disappears after treatment. Patients with adenoid cystic carcinoma who have a complete response (CR) or partial response (PR) per RECIST criteria v. 1.1 will be included in the results. Per RECIST v. 1.1, CR is defined as "disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm." A PR is defined as "At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters."
Time Frame: On Cycle 2 Day 1, and every cycle thereafter (1 cycle = 12 weeks), about 27 months
Population: Adenoid Cystic Carcinoma (ACC) patient only.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 18
percent of participants | .06 [0.01 to .26]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) is defined as the percentage of patients with Complete Response (CR), Partial Response (PR), and Stable Disease (SD) and will be assessed by RECIST 1.1 in patients with adenoid cystic carcinoma (ACC). Per RECIST v. 1.1, CR is defined as, "Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm." PR is defined as, "At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters." SD is defined as, "Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study."
Time Frame: On Cycle 2 Day 1, and every cycle thereafter (1 cycle = 12 weeks), about 27 months
Population: Patients with Adenoid cystic carcinoma only.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 18
percent of participants | 0.71 [0.47 to .87]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as time in months from the date of first study treatment to the date of death or withdrawal from study, whichever comes first. The percentage of patients alive at 6 months, 12 months, and 24 months will be reported. All patients who receive at least one dose of nivolumab will be included in the secondary analyses of OS.
Time Frame: Up to 2 years from start of treatment
Population: Patients with Adenoid Cystic Carcinoma only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 19
percentage of participants
  Overall Survival at 6 months | 89.47 [76.69 to 100]
  Overall Survival at 12 months | 73.68 [56.32 to 96.4]

6. Secondary Outcome: Number of Adverse Events Possibly Related to Study Drugs Graded 3, 4, and 5
Description: Toxicity, both frequency and severity, will continue to be measured by monitoring the occurrence of adverse events. Adverse events will be defined as those included in CTCAE v 4.03. AEs that were determined to be at least possibly related to study drug and graded 3, 4, 5 are included here. Grade 1 (mild): the event causes discomfort without disruption of normal daily activities. Grade 2 (moderate): the event causes discomfort that affects normal daily activities. Grade 3 (severe): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status. Grade 4 (Life-threatening): the patient was at risk of death at the time of the event. Grade 5 (fatal): the event caused death.
Time Frame: Up to 30 days after discontinuation, where range of cycles attempted was 1-11, where 1 Cycle = 84 days/12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 24
Participants
  Fatigue | 1
  Lymphocyte Count Decreased | 4
  Anemia | 2
  Aspartate Aminotransferase increased | 1
  Diarrhea | 1
  Anorexia | 1
  Alanine Aminotransferase Increased | 1
  Weight Loss | 1
  Adrenal Insufficiency | 1
  Rash maculo-papular | 1
  Alkaline Phosphatase Increased | 1
  Colitis | 1
  Mucositis oral | 1
  Hypokalemia | 1
  Hypophosphatemia | 1
  Serum Amylase Increased | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 3 year period, and is still continuing (2 patients still on treatment). For other AEs, each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment. For Serious AEs, each patient was followed at time of consent and 100 days post last treatment. 1 Cycle = 84 days/12 weeks and the range of cycles attempted was 1-11.
Description: A patient who was registered and signed consent but did not initiate treatment is included as at risk for SAE but not at risk for other AEs. This patient never received treatment on study. All cause mortality and other adverse events are assessed from first dose of study treatment. Only patients that received at least 1 dose of study drug are included in all cause mortality and other adverse events. SAEs are assessed from patient signing consent.
Arm/Group | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 11/24
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=25)
Spinal fracture (Injury, poisoning and procedural complications) | 1 — The patient also experienced tumor pain at the time of this event.
ascites (Gastrointestinal disorders) | 1 — The patient also experienced increased blood bilirubin and cholecystitis at the time of this event.
fever (General disorders) | 1
sinusitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1 — The patient also experienced an increase in Aspartate aminotransferase at the time of this event.
Neck pain (Musculoskeletal and connective tissue disorders) | 1
nausea (Gastrointestinal disorders) | 1 — The patient also experienced constipation at the time of this event.
Colitis (Gastrointestinal disorders) | 2 — One patient also experienced nausea and diarrhea at the time of this event.
Thromboembolic event (Vascular disorders) | 2
acute kidney injury (Renal and urinary disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 — The patient also experienced acute kidney injury and alkalosis at the time of this event.
Pain Right Lower Limb (Musculoskeletal and connective tissue disorders) | 1 — The patient also experienced muscle weakness in the right lower limb at the time of this event.
Adrenal Insufficiency (Endocrine disorders) | 2 — The patient also experienced anorexia at the time of this event.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Adenoid Cystic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
anorexia (Metabolism and nutrition disorders) | 1 — The patient also experienced hypotension at the time of this event.
Port Malfunction (Injury, poisoning and procedural complications) | 1
Viral Gastroenteritis (Gastrointestinal disorders) | 1 — The patient also experienced a respiratory infection (possible pneumonia) at the time of this event.
confusion (Psychiatric disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Anxiety (Psychiatric disorders) | 1 — The patient also experienced fatigue and pain in the chest wall at the time of this event.
Abdominal Pain (Gastrointestinal disorders) | 1 — The patient also experienced non-cardiac chest pain at the time of this event.
sepsis (Infections and infestations) | 1 — The patient also experienced non-cardiac chest pain, dyspnea, anorexia, and respiratory failure at the time of this event.
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 — One patient also experienced abdominal pain at the time of this event. One patient also experienced pericardial effusion and sepsis at the time of this event. One patient also experienced pain at the time of this event.
headache (Nervous system disorders) | 1
Left Jaw Cellulitis (Skin and subcutaneous tissue disorders) | 1 — One patient also experienced left jaw cellulitis at the time of this event.
seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=24)
Abdominal pain (Gastrointestinal disorders) | 3
Adrenal insufficiency (Endocrine disorders) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 10
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Amnesia (Nervous system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 15
Anisocoria (Eye disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3
bilateral temporal bulging (Nervous system disorders) | 1
Blood bilirubin increased (Investigations) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Cachexia (General disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Chronic erythematous rash (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Creatinine increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
desquamation (Skin and subcutaneous tissue disorders) | 1
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
edema of c-spine (General disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Epigastric burning (Gastrointestinal disorders) | 1
erythema (Skin and subcutaneous tissue disorders) | 1
erythema in throat (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 12
Fibrinogen decreased (Investigations) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (General disorders) | 2
Flushing (Vascular disorders) | 1
Gait disturbance (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 4
Hearing impaired (Ear and labyrinth disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 20
Hyperthyroidism (Endocrine disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophonia (Musculoskeletal and connective tissue disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 7
Infusion related reaction (General disorders) | 1
INR increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Left facial droop (General disorders) | 1
Left facial paralysis (General disorders) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 17
Mucositis oral (Gastrointestinal disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Non-cardiac chest pain (General disorders) | 2
Numbness/ pain forearm (Musculoskeletal and connective tissue disorders) | 1
Numbness/ tingling of the arm (General disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Platelet count decreased (Investigations) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Respiratory, thoracic and mediastinal disorders - NOS (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (General disorders) | 1
Right arm pain/ weakness (General disorders) | 1
Right hand atrophy (Musculoskeletal and connective tissue disorders) | 1
Right lower eyelid stye (Eye disorders) | 1
Sensation of Thick Tongue (Investigations) | 1
Serum amylase increased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Somnolence (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tremor (Nervous system disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 1
Urine output decreased (Investigations) | 1
Visual changes (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 3
Weight loss (Investigations) | 11
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study closed without meeting the total accrual goal due to contract issues with the pharma company.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03146650/Prot_SAP_000.pdf